CLINICAL TRIAL: NCT03445884
Title: 68Ga-NODAGA-E[c(RGDγK)]2: a Novel Positron Emission Tomography (PET) Tracer for in Vivo Molecular Imaging of Myocardial Angiogenesis Following Myocardial Infarction
Brief Title: 68 Ga-NODAGA-E[c(RGDγK)]2: Positron Emission Tomography Tracer for Imaging of Myocardial Angiogenesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Simon Bentsen, Medical Doctor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUDRACR-number: 2017-002709-36
Record Dates: First submitted 2018-02-18; First posted 2018-02-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Acute Myocardial Infarction
Keywords: positron emission tomography; nuclear medicine; prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute myocardial infarctions group (Experimental): 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV. three times. 1-3 days after intervention, 7-10 days after intervention and 30-35 days after intervention.
  Interventions: Drug: 68Ga-NODAGA-E[c(RGDyK)]2
- Control group (Active Comparator): 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV. one time.
  Interventions: Drug: 68Ga-NODAGA-E[c(RGDyK)]2

INTERVENTIONS:
Drug: 68Ga-NODAGA-E[c(RGDyK)]2 — 200 MBq 68Ga-NODAGA-E[c(RGDyK)]2 administered IV.
  Other Names: RGD-PET

SUMMARY:
The aim is to examine the expression of αvβ3 integrin using a novel selective radiotracer in patients with myocardial infarction and investigate if it is a suitable tool for predicting myocardial recovery and thus prognosis.

DETAILED DESCRIPTION:
Ischemic heart disease is worldwide the single most frequent cause of death. The number of patients surviving acute myocardial injury is increasing due to improved acute treatment. However, after the initial repair, the tissue undergoes a remodeling phase to compensate for the damaged area. This re-modeling phase can change the structure end geometry of the heart resulting in lower ejection fraction, leading to cardiac dysfunction, which eventually leads to heart failure. Understanding and ideally modifying the reparative mechanisms following myocardial infarction is increasingly important and may lead to improved outcome.

If the heart suffers from ischemia following an acute coronary event, the tissue reacts strongly to the hypoxia. The body will as a compensatory mechanism create new vessel to provide the tissue with oxygen. This is known as the biological process of angiogenesis. This complex process involves different angiogenic and pro-fibrotic transcription factors that initiate the restoration of capillaries by sprouting from the existing endothelial cells in response to hypoxia.

Time seem essential to protect and save the myocardium. An early onset of cytokines and growth factors is associated with a decline in cardiomyocytes apoptosis, smaller infarct areas, and decreased ventricular dilation. Therefore, an early induction of angiogenesis seems important for a good prognosis of the patient.

Integrin αvβ3 is a transmembrane cell surface receptor that is markedly upregulated in states of angiogenesis. It facilitates migration and proliferation and thereby allowing cells to respond to extracellular environment. Integrin αvβ3 is thus a key player in the angiogenic process. The integrin αvβ3 has a binding site for an RGD peptide (Arg-Gly-Asp motif) and this can be targeted by PET tracers.

RGD-based PET tracers have been shown to accumulate at the site of myocardial necrosis in both human and animal studies. The uptake seems to peak a few weeks after the infarction and may correlate to recovery of cardiac function and thus serve as a prognostic marker.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years

Acute myocardial infarction Group:

* Verified first-time acute myocardial infarction treated with PCI

Control Group:

* Previous healthy
* No known cardiac disease

Exclusion Criteria:

* No prior history of acute coronary infarction
* No prior history of Heart surgery
* Not treated with anti-angiogenic medicine
* Subject with pacemaker, cochlear implant or insulin pump
* Pregnancy
* Lactation
* Severe claustrophobia
* Severe obesity (weight above 140kg)
* If a subject is in the fertile age, a pregnancy test will be use prior to injection to the PET_tracer
* If a subject is having a severe allergic reaction to the PET-tracer, the person will be excluded for the rest of the trial
* If the PET-tracer is administered subcutaneous, the person will be excluded for the rest of the trial¨
* Tupe I or II diabetes

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate myocardial angiogenesis | 30-35 days
  Analysing uptake of 68Ga-NODAGA-E[c(RGDyK)]2 Positron Emission Tomography in myocardial infarction after PCI

SECONDARY OUTCOMES:
Uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and myocardial perfusion | 30-35 days
  Quantitative uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and change in myocardial perfusion after PCI using Rubidium 82 Positron Emission Tomography after Percutaneous coronary intervention(PCI)
Uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and functional recovery | 30-35 days
  Quantitative uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and functional recovery using Magnetic Resonance after PCI
Uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and viability | 30-35 days
  Quantitative uptake of 68Ga-NODAGA-E[c(RGDyK)]2 and viability using Flour-Deoxy-Glucose Positron Emission Tomography after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Department of Physiology, Nuclear Medicine and PET, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No